CLINICAL TRIAL: NCT07205744
Title: Management of Post-Menopausal Skin Complaints: An Open Label Study
Brief Title: Post-Menopause Skin Rejuvenation Study
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Erevna Innovations Inc. (Other)
Responsible Party: Principal Investigator, Andreas Nikolis, Principal Investigator, MD, PhD, Erevna Innovations Inc.
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GAL-2025-MENO-75
Record Dates: First submitted 2025-09-18; First posted 2025-10-03 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Aesthetic; Menopause; Post-menopause; Injectables; Biostimulator; Hyaluronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primary Complaint: Lack of skin hydration (Other): Participants presenting with a primary complaint of lack of skin hydration will be administer primarily with Restylane SkinBoosters Vital followed by Sulptra Aesthetic
  Interventions: Device: Restylane SkinBoosters Vital
- Primary Complaint: Loss of skin elasticity (Other): Participants presenting with a primary complaint of lack of skin elasticity will be administer primarily with Sculptra Aesthetic followed by Restylane SkinBoosters Vital
  Interventions: Drug: Sculptra Aesthetic

INTERVENTIONS:
Device: Restylane SkinBoosters Vital — Restylane® Skinboosters™ Vital (HASBV) is manufactured by Galderma Laboratories. It is a sterile non-animal hyaluronic acid (20mg/mL) based gel that is supplied in a 1mL glass syringe. The syringed is packed with a 29G TW (thin-walled) needle.
  For this study, commercial products will be used. The study products are for single use only.
  Arms: Primary Complaint: Lack of skin hydration
Drug: Sculptra Aesthetic — Sculptra® Aesthetic (PLLA-SCA) is manufactured by Galderma Laboratories. It is a sterile, lyophilized preparation of PLLA that is biocompatible and biodegradable. Each vial contains 367.5 mg of freeze-dried powder, including 150 mg of PLLA. Prior to injection, it will be reconstituted with sterile water for injection (SWFI) and lidocaine hydrochloride (2%).
  For this study, commercial products will be used. The study products are for single use only.
  Arms: Primary Complaint: Loss of skin elasticity

SUMMARY:
The post-menopausal state is marked by a sharp decline in estrogen, leading to significant structural and functional changes in the skin, including collagen loss, dryness, thinning, and reduced elasticity. To address these concerns, aesthetic injectables products such as Sculptra® Aesthetic (poly-L-lactic-acid [PLLA- SCA]) and Restylane Skinboosters®[HASBV] (small-particle hyaluronic acid - SP-HA) can be used. PLLA-SCA stimulates collagen production via cellular activation (biostimulator), gradually improving dermal structure. HASBV enhances hydration, elasticity, and skin texture when injected under the skin.

Considering that hydration and laxity represent the primary aesthetic concerns in this patient population. Targeted treatment with SP-HA (HASBV) to improve hydration and PLLA-SCA to address laxity have been shown to produce significant clinical outcomes by directly addressing these key dermal deficiencies. This approach forms the basis of the current study.

DETAILED DESCRIPTION:
This study is a prospective, controlled, open-label study involving fifty (50) post-menopausal adult female participants between the age of 40 and 65, who are both utilizing and not utilizing Hormone Replacement Therapy (HRT) to control post-menopausal symptoms. All participants with facial or décolleté skin aging will be considered eligible for treatment following completion of the informed consent process and Baseline evaluation.

Randomization (as primary participant complaint) will be undertaken to allocate participants to one of two groups:

* Group A (Hydration as Primary Complaint): HASBV followed by PLLA-SCA (n = 25)
* Group B (Laxity as Primary Complaint): PLLA-SCA followed by HASBV (n = 25)

ELIGIBILITY:
Inclusion Criteria:

1. Participants must voluntarily sign and date an informed consent, approved by an independent ethics committee, prior to the initiation of any screening or study-specific procedures.
2. post-menopausal participants between the age of 40 and 65 years old;
3. Participants with a -menopausal status (at least 12 consecutive months of amenorrhea without other pathological or physiological causes).

   • A clinical evaluation will be undertaken by a clinical professional to determine post-menopausal status.
4. Participants with established clinical signs of skin aging including but not limited to: reduced skin elasticity, increased wrinkling, dryness, volume loss and/or contour deficits.
5. Participant is willing and able to comply with procedures required in the protocol.
6. Participant must be in good health as per investigator's judgment based on medical history
7. For subgroup analysis: either currently on stable-dose HRT for ≥ 6 months or not receiving any form of HRT for ≥6 months

Exclusion Criteria:

1. Previous biostimulators 18 months prior to this study;
2. Previous SP-HA 18 months prior to this study;
3. Previous HA injectables 18 months prior to study in the facial and décolleté region;
4. Participant has an uncontrolled systemic disease.
5. Participant presents with or has a history of any medical condition that may place the participant at an increased risk following exposure to hyaluronic acid or interfere with the study evaluation, including:

   * Diagnosed myasthenia gravis, Lambert-Eaton syndrome, amyotrophic lateral sclerosis, or any other significant disease that might interfere with neuromuscular function
   * History of facial nerve palsy
   * Infection or dermatological condition at the treatment injection sites
   * Marked dermatochalasis, deep dermal scarring, excessively thick sebaceous skin, or excessively photodamaged skin
6. Participant has a history of clinically significant medical conditions or any other reason that the investigator determines would interfere with the participant's participation in this study or would make the participant an unsuitable candidate to receive the study medical device.
7. Participant has a history of an allergic reaction or significant sensitivity to constituents of the study medical device (or its excipients) including Vicryl
8. Participant has an tattoos, jewellery, or clothing which obscure the treatment area and cannot be removed.
9. Participant has an anticipated need for surgery or overnight hospitalization during the study.
10. Participant has a history of surgical procedures in intended treatment areas, including any lifting procedure (e.g., facial lift, suture lift, thread lift, brow lift, eyelid and/or eyebrow surgery, neck lift).
11. Participant with known active COVID infection within 14 days of baseline treatment.
12. Participant is currently enrolled in another clinical study.
13. Participant is presenting with porphyria.
14. Participant presents with active disease, such as inflammation, infection or tumors, in or near the intended treatment sites.
15. Participant has a bleeding disorder or take thrombolytics or anticoagulants.
16. Participant has a need to take immunosuppressants.
17. Participant has undergone dental procedures including teeth cleaning withing 14 days prior to baseline treatment
18. Participant has undergone any vaccine administration withing the 14 days prior to treatment administration
19. Participant categorised as a heavy smoker, more than 12 cigarettes per day

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2025-08-14 (Actual); Primary Completion 2026-08-28 (Estimated); Study Completion 2026-09-28 (Estimated)

PRIMARY OUTCOMES:
Evaluate the efficacy of HASBV and PLLA-SCA in improving skin-related clinical outcomes in the post-menopausal population. | Baseline to Week 26
  Frequency of participants having at least "improved" (e.g., "improved", "much improved" or "very much improved") on the Global Aesthetics Improvement Scale (GAIS) of the face and décolleté regions, as graded by a blinded evaluator with two-dimensional and/or three-dimensional (2D and 3D) photography, at all visits (Canon EOS, VISIA, Canfield Scientific).

SECONDARY OUTCOMES:
Evaluate the impact of HASBV and PLLA-SCA treatments on facial skin in the post-menopausal population using Objective Parameters | Baseline to Week 36
  Assess changes in skin parameters using the Courage+Khazaka electronic GmbH instrumentation
Evaluate the impact of HASBV and PLLA-SCA treatments on facial skin in the post-menopausal population using Histological analysis of treated skin in a subset of consenting participants | Baseline, Week 12-16, Week 28-36
  Assess changes in biological parameters in tissue samples from baseline
Evaluate the impact of HASBV and PLLA-SCA treatments on the décolleté skin in the post-menopausal population using: Objective Parameters | Baseline Week 36
  Changes in Skin parameters using the Courage+Khazaka electronic GmbH instrumentation
Evaluate participants satisfaction with the treatment regimen for the face and décolleté. | Week 4-6 to Week 36
  Proportion of Participants being at least satisfied ("satisfied", "very much satisfied", or "extremely satisfied") with treatment at all visits after baseline (Visit 2 to Visit 8),using the seven-point participant satisfaction with treatment questionnaire.

OTHER OUTCOMES:
Subgroup Analysis of Treatment Response Between HRT-Treated and Non-HRT-Treated Post-Menopausal Participants | Baseline to Week 36
  Comparison of treatment response to HASBV and PLLA-SCA regimens between HRT-treated and non-HRT-treated post-menopausal participants using appropriate statistical methods.
Change in Facial and Décolleté Skin Thickness using high frequency ultrasonography | Baseline to Week 36
  Measurement of skin thickness changes from baseline using ultra-high-frequency ultrasound (Clarius L20 HD3, BC, Canada) in facial and décolleté regions following treatment with HASBV and PLLA-SCA.
Incidence and Severity of Adverse Events (AEs) | Baseline to Week 36
  Frequency and severity of physician-reported and participant-reported adverse events throughout the study duration.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Nikolis, MD, PhD, Principal Investigator — Erevna Innovations Inc.
Locations (1):
- Erevna Innovations Inc., Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No